CLINICAL TRIAL: NCT01291797
Title: Use of AEEG as Predictor of Long-term Motor Outcome in Neonates With Congenital Heart Disease
Status: Terminated | Type: Observational
Why Stopped: due to inability to recruit sufficient sample size in reasonable time frame.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Ian Holzman, MD, Principal Investigator, Mount Sinai Hospital Division of Newborn Medicine
Other Study IDs: MSSM 10-0568
Record Dates: First submitted 2011-02-03; First posted 2011-02-08 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease; neurodevelopmental outcome; AEEG; sleep wake cycles
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonates with congenital heart disease: The case group will consist of newborns born between 32 and 41 weeks gestation diagnosed with a congenital cardiac anomaly requiring surgical repair during their hospitalization and managed in the Mount Sinai Neonatal Intensive Care Unit. The control arm will include newborns born between 32 and 41 weeks without congenital cardiac anomalies. Both groups will undergo a neurological screening assessment and receive an AEEG to look at sleep wake cycles.

SUMMARY:
This study aims to examine performance on a neurological screening test, the Dubowitz, and sleep wake cycles on amplitude integrated electroencephalogram (AEEG) in neonates with congenital heart disease (CHD) as a way to potentially predict longterm motor outcome. It will compare the results of these studies to neonates without CHD.

DETAILED DESCRIPTION:
Neonates with congenital heart disease are at increased risk of adverse long term neurodevelopmental outcomes, including lower mean intelligent quotients (IQs). However, it is difficult to predict with neonates are most likely to be affected and a cost effective method is needed. AEEG has been used in neonates with hypoxic-ischemic encephalopathy and abnormal sleep wake cycles have been proposed to predict poorer long term outcomes. We thus hypothesize that abnormal sleep wake cycles in neonates with congenital heart disease will correlate with poorer outcomes. In our study, we will examine the relationship between performance on a neurodevelopmental screening tool, the Dubowitz neonatal neurological screening tool, and the sleep wake cycles on AEEG both before and after cardiac repair to try and predict which neonates are at increased risk of adverse long term outcomes. We will also compare the findings of the AEEG and performance on the neurodevelopmental tool to the data gathered from neonates without cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Newborn with cardiac anomaly requiring surgical intervention or a newborn that is in NICU for at least 24 hours for monitoring
* If newborn has congenital cardiac anomaly, cardiac repair must be performed at Mount Sinai Hospital
* If newborn has congenital cardiac anomaly, he/she must be managed pre-operatively for at least 24 hours at Mount Sinai Hospital
* If newborn has congenital cardiac anomaly, he/she must be managed post-operatively at Mount Sinai Hospital for at least 72 hours

Exclusion Criteria:

* Newborns with previously known anomalies other than cardiac
* Chromosomal abnormalities other than 22Q, that might have long-term neurodevelopmental implications
* Diagnosis of hypoxic-ischemic encephalopathy
* Metabolic disorder
* Other genetic disorders

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Anticipated, 65 newborns with congenital heart disease and 20 newborns without congenital heart disease
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Abnormal sleep wake cycles on AEEG | from 24 hours of life to time of discharge home from the neonatal intensive care unit (NICU) which is on average about four weeks

SECONDARY OUTCOMES:
Performance on neurologic screening tools | from 24 hours of life to time of discharge home from the neonatal intensive care unit which is on average about four weeks
Head ultrasound abnormalities | from 24 hours of life to time of discharge home from the neonatal intensive care unit which is on average about four weeks
Seizures | from 24 hours of life to time of discharge home from the neonatal intensive care unit which is on average about four weeks
Death | from 24 hours of life to time of discharge home from the neonatal intensive care unit which is on average about four weeks
Inability to feed orally | from 24 hours of life to time of discharge home from the neonatal intensive care unit which is on average about four weeks
Respiratory support requirement | from 24 hours of life to time of discharge home from the neonatal intensive care unit which is on average about four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian Holzman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital Division of Newborn Medicine, New York, New York, United States

REFERENCES:
- [Background] Massaro AN, El-Dib M, Glass P, Aly H. Factors associated with adverse neurodevelopmental outcomes in infants with congenital heart disease. Brain Dev. 2008 Aug;30(7):437-46. doi: 10.1016/j.braindev.2007.12.013. Epub 2008 Feb 4. PMID 18249516
- [Background] Brown MD, Wernovsky G, Mussatto KA, Berger S. Long-term and developmental outcomes of children with complex congenital heart disease. Clin Perinatol. 2005 Dec;32(4):1043-57, xi. doi: 10.1016/j.clp.2005.09.008. PMID 16325677
- [Background] Limperopoulos C, Majnemer A, Shevell MI, Rosenblatt B, Rohlicek C, Tchervenkov C. Neurodevelopmental status of newborns and infants with congenital heart defects before and after open heart surgery. J Pediatr. 2000 Nov;137(5):638-45. doi: 10.1067/mpd.2000.109152. PMID 11060529
- [Background] Shalak LF, Laptook AR, Velaphi SC, Perlman JM. Amplitude-integrated electroencephalography coupled with an early neurologic examination enhances prediction of term infants at risk for persistent encephalopathy. Pediatrics. 2003 Feb;111(2):351-7. doi: 10.1542/peds.111.2.351. PMID 12563063